CLINICAL TRIAL: NCT02732808
Title: Evaluation of Outcome of Double Stimulation and Egg Collection in the Same IVF/ ICSI Cycle in Poor Ovarian Responders
Brief Title: Dual Ovarian Stimulation in the Same IVF/ICSI Cycles for Treatment of Poor Ovarian Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-022
Record Dates: First submitted 2015-07-07; First posted 2016-04-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: Double stimulations; luteal-phase ovarian stimulation; poor ovarian response
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- poor ovarian responder (Experimental): The women with diagnose of poor ovarian responder after IVF/ICSI treatments underwent ovulation stimulation and egg collection in the same IVF/ ICSI cycle ( Shanghai protocol)
  Interventions: Drug: Ovulation stimulation

INTERVENTIONS:
Drug: Ovulation stimulation — Double stimulation in 2 phases:
  Phase I: Clomiphene citrate (Ovumid®) 25 mg/day with co-treatment of Letrozole (Letrofem®) 2.5 mg/day are given from cycle day 3 onwards. Letrozole (Letrofem®) 2.5 mg/day are given from cycle day 3 onwards. human menopausal gonadotrophin (HMG) Menopur®150 IU every other day beginning on cycle day 6. triptorelin (Decapeptyl®) 100 μg follows by ibuprofen 600 mg.
  Phase 2:A total of 225 IU HMG(Decapeptyl®) and letrozole (Letrofem®) 2.5 mg is administered daily .Daily administration of medroxyprogesterone acetate (Progestrone®)10 mg. . the final stage of oocyte maturation is induced again with triptorelin (Decapeptyl®)100 μg by injection.

SUMMARY:
This study is a prospective before & after clinical trial to investigate the efficacy of double stimulations during both the follicular and luteal phases in patients with poor ovarian response undergoing IVF and intracytoplasmic sperm injection (ICSI) cycles.

The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute. The study is conducted according to the Declaration of Helsinki for medical research. All participants provide informed consent after counseling for infertility treatments and routine IVF/ICSI programs.

All the patients who diagnosed as poor ovarian responders (POR) based on the Bologna criteria are eligible for participation in this study. In order to define the poor response in IVF, at least two of the following three features must be present: (i) advanced maternal age or any other risk factor for POR; (ii) a previous POR; and (iii) an abnormal ovarian reserve test (ORT). Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT.

Stage one of treatment protocol First stimulation performs by Clomiphene citrate (Ovumid®, Iran Hormones Company) 25 mg/day with co-treatment of Letrozole (Letrofem®, Iran Hormones Company) 2.5 mg/day are given from cycle day 3 onwards. Letrozole is only given for 4 days and clomiphene citrate is continuously used before the trigger day. Patients start to inject human menopausal gonadotrophin (HMG) (Menopur®, Ferring, Switzerland) 150 IU every other day beginning on cycle day 6. When one or two dominant follicles (18 mm in diameter) observed, the final stage of oocyte maturation will be induced with triptorelin 100 μg (Decapeptyl®; Ferring GmbH, Germany) follows by ibuprofen 600 mg (Ibuprofen-Najo® , Coated Tablets, Najo Company, Iran) is used on the day of oocyte maturation triggering and the day after. After the first oocyte retrieval, human menopausal gonadotrophin and letrozole are administrated to stimulate follicle development, and oocyte retrieval will be carried out a second time when dominant follicles have matured. All highest-quality embryos (including grade 1 and grade 2, eight-cell blastomere embryos) will be cryopreserved by vitrification method on the third day after oocyte retrieval.

Stage two of treatment protocol:

Transvaginal ultrasound evaluation performs after oocyte retrieval to determine whether to continue the second ovarian stimulation. The criterion for continued stimulation is the presence of at least two antral follicles 2-8 mm in diameter. A total of 225 IU HMG (Menopur®, Ferring, Switzerland) and letrozole 2.5 mg (Letrofem®, Iran Hormones Company) is administered daily from the day of, or the day after, oocyte retrieval. The initial second stage follicular monitoring is conducted 5-7 days later, and then for follow up every 2-4 days, by using a transvaginal ultrasound evaluation, to record the number of developing follicles. Letrozole administration is discontinued when the dominant follicles reached diameters of 12 mm, given that large follicles have redundant LH and FSH receptors, and good response to exogenous hormone stimulations. Daily administration of medroxyprogesterone acetate 10 mg (Progestrone®, 5mg bid; Aboureihan, Iran) is added beginning on stimulation day 12 for cases in which post-ovulation follicle size is smaller than 14 mm in diameter and stimulation needed to continue for several more days. This performs to postpone menstruation and avoid oocyte retrieval during menstruation, to prevent the risk of infection from the procedure. When three dominant follicles reached diameters of 18 mm or one mature dominant follicle exceeded 20 mm, the final stage of oocyte maturation is induced again with triptorelin 100 μg (Decapeptyl®; Ferring GmbH, Germany) by injection. Again, ibuprofen 600 mg (Ibuprofen-Najo® , Coated Tablets, Najo Company, Iran) is used on the day of oocyte maturation triggering and the day after. Transvaginal ultrasound-guided oocyte retrieval was conducted 32-36 h after GnRH agonist administration. All retrieved oocytes were treated same as in the study stage one.

DETAILED DESCRIPTION:
Data collection will be performed by using questionnaire to be filled as per the available records and laboratory results. The mean of total number of retrieved oocytes and embryos after the present protocol were compared with the mean of total number of retrieved oocytes and embryos at previous routine cycle.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Poor ovarian response (POR), according to Bologna criteria:

the patients have at least two of the following criteria:

* age over 40 years;
* a history of ovarian surgery;
* previous treatment using conventional protocols that yielded less than three oocytes;
* antral follicle count of less than 5 on menstrual cycle day 2-3; and basal serum Follicle Stimulating Hormone ( FSH) concentration between 10 and 19 IU/l.

Exclusion Criteria:

* ovarian failure including basal Follicle Stimulating Hormone ( FSH) above 20 IU/l or no antral follicle by ultrasound examination;
* Endometriosis grade 3 or higher;
* Any contraindications to ovarian stimulation treatment.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | 32-36 hours
  Evaluation the Total number of retrieved oocytes 32- 36 hours after Gonadotropin Releasing Hormone (GnRH )agonist injection.

SECONDARY OUTCOMES:
Quality of obtained embryos | 3 days after oocyte retrieval
  we score embryo quality according to the following quality criteria: Excellent (Day 3: 6-8 even size blastomeres with ≤10% fragmentation), Good (Day 3: 6-8 even or uneven size blastomeres with 10%-20% fragmentation), Poor (Uneven and few blastomeres with >20% fragmen¬tation).

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran; Mandana Hemmat, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Arezoo Arabipoor, MSc, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org